CLINICAL TRIAL: NCT06214065
Title: Modulating Temporoparietal Junction Mentalizing-Related Activity in Autism Spectrum Disorder Using Transcranial Magnetic Stimulation
Brief Title: Modulating Temporoparietal Junction Mentalizing-Related Activity in Autism Spectrum Disorder (ASD) Using Transcranial Magnetic Stimulation (TMS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HHC-2023-0203; R01MH132044 (NIH); Assaf 121223 (Other: Yale); 2000039667 (Other: Yale IRB)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ASD: excitatory, then inhibitory, then sham rTMS (Experimental): Participants in this group will undergo fMRI pre- and post- rTMS. Each will receive an excitatory, inhibitory and sham rTMS to the right temporoparietal junction (TPJ) on mentalizing task-related (MTR) activity over 4 study visits.
  Interventions: Diagnostic Test: fMRI; Device: rTMS
- Typically Developing (TD): excitatory, then inhibitory, then sham rTMS (Experimental): Participants in this group will undergo fMRI pre- and post- rTMS. Each will receive an excitatory, inhibitory and sham rTMS to the right temporoparietal junction (TPJ) on mentalizing task-related (MTR) activity over 4 study visits.
  Interventions: Diagnostic Test: fMRI; Device: rTMS

INTERVENTIONS:
Diagnostic Test: fMRI — fMRI will be performed pre- and post-rTMS
Device: rTMS — TMS procedures are scheduled during study sessions 2-4 between the two MRI scans on those days. Because rTMS induces neural changes that last about 1 hour, rTMS will be applied immediately before the second MRI scan on each day. Prior to the TMS visits, target coordinates and orientation vectors will be generated from the MRI data and the e-field models and loaded into Localite along with the participant's reconstructed T1 image. During the visits, the participant's head will be co-registered to the T1 using fiducial points at the Nasion and Tragi. TMS pulses will be delivered, using the Localite software to target and track the optimal orientation calculated with e-field modeling.

SUMMARY:
The goal of this observational study is to test the modulation effect of different transcranial magnetic stimulation (TMS) on the neural network supporting our ability to create mental representations of others (also known as mentalizing) in young adults with autism. The main question it aims to answers is can stimulation of the right temporoparietal junction can change brain activity related to mentalizing during social interaction in the stimulation area and other brain areas connected to it. Researchers will compare results to a group of individuals without autism to see if the patterns of neural activity change are similar between the groups.

Participants will undergo assessment of their clinical traits and social skills and baseline MRI scan. They will attend three additional visits that include TMS session and functional MRI scans before and right after TMS.

DETAILED DESCRIPTION:
All participants will be scheduled for four study sessions that include a baseline and three subsequent sessions that will each include two functional magnetic resonance imaging (fMRI) scans, one pre and one post an rTMS session.

During each fMRI scan, participants will be engaged in intersocial, competitive Domino task that involves mentalizing. rTMS manipulation, administered in a double-blind, counterbalanced fashion, includes one session each of excitatory (intermittent theta-burst stimulation, iTBS), inhibitory (continuous TBS, cTBS), and sham sequences. The rTMS will be guided with individualized electric-field modeling calculated from a structural MRI scan collected on the baseline session. This robust design is necessary to identify the optimal rTMS sequence to engage the right TPJ and the mentalizing network in ASD because firm conclusions about how best to modulate this network cannot be drawn from the few known published reports.

Investigators hypothesize that iTBS will result in increased, while cTBS in decreased MTR neural activity in the mentalizing network, with this being more pronounced in ASD, and sham resulting in no change. Understanding this mechanism will be the first and crucial step in validating rTMS of the right TPJ as a viable neural target to modulate neural circuit, and subsequently to modulate social-communication skills in ASD in future clinical studies. The significance of such a line of research should be considered in the context of the high prevalence of ASD and the dire need of developing effective interventions, especially for adults.

The three rTMS sessions will be compared within-subject and between-groups.

ELIGIBILITY:
Inclusion Criteria:

* Estimated full-scale IQ>80
* Right handed
* Fluent in English
* Individual can cooperate with all study's procedures
* No history of neurological disorder (e.g. epilepsy) or neurosurgery
* No major medical condition (e.g. cancer, heart failure)
* No history of significant head injury
* No primary relatives with history of any neurological disorder with a potentially hereditary basis, including epilepsy or MS
* No current use of medications with psychotropic (e.g., benzodiazepines) or anti- or pro-convulsants
* No current substance use (determined by urine screen and breathalyzer in all visits)
* Negative urine pregnancy (women) test at time of MRI scans
* No MR contra-indications (e.g. in-body metal implant, severe claustrophobia)
* No previous participation in our lab in a study including the Domino fMRI task
* For ASD: Stable medication treatment 4 weeks prior to study enrollment
* For Control Group: No current or history of psychiatric disorders, other than simple phobia, and/or primary relatives with ASD

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mentalizing Task Related (MTR) neural activity in the mentalizing network | during each fMRI, up to 5 hours
  Change in MTR activity in six brain regions, from fMRI scans will be measured pre- to post-rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Vaughn Steele, MD, Principal Investigator — Yale University; Michal Assaf, MD, Principal Investigator — Yale University
Locations (1):
- Olin Neuropsychiatry Research Center (ONRC), Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All investigators are aware of and agree to abide by the principles for sharing research resources, as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs." Specifically, all data collected in this study, including demographic information, psychiatric, symptom, cognitive and social assessments as well as MRI imaging data, will be shared with the scientific community through the National Institute of Mental Health Data Archive (NDA).
Access Criteria: National Institute of Mental Health Data Archive (NDA)